CLINICAL TRIAL: NCT00831168
Title: The Bliss Cluster Randomised Control Trial on the Effects of Active Dissemination of Information on Outcomes of Premature Babies.
Brief Title: BEADI - The Bliss Cluster Randomised Control Trial on the Effects of Active Dissemination of Information (BEADI)
Acronym: BEADI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Confidential Enquiry into Maternal and Child Health (Other)
Responsible Party: Richard Congdon, CEMACH
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BEADI2005
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Premature Babies
Keywords: neonatal; premature babies; healthcare research; Babies born before 27 weeks gestation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Effects of Active Dissemination — No medical intervention involved. It is purely information based.

SUMMARY:
BEADI is a dissemination trial, on standards of care of premature babies. The main objective of BEADI is to assess whether an innovative 'active' strategy for the dissemination of neonatal information (evidence reviews, interactive training workshop, benchmarking and feedback, and ongoing support) is more likely to lead to changes in policy and practice than the traditional (more passive) forms of dissemination in English neonatal units.

BEADI will focus on three areas of neonatal care for premature (22+0 to 26+6 weeks' gestation) babies born in England: timing of surfactant therapy, staffing for resuscitation at delivery, and temperature control (in line with the main Project 27/28 findings ). However, the approach is applicable to a wide variety of clinical policies and practice.

The BEADI study has been granted ethical approval by MREC to use a subset of data collected by EPICure2 up until 31st December 2006 (pre-intervention data). For the post-intervention data, ethical approval has been granted for CEMACH to continue data collection against the three clinical areas using a subset of data items captured in the PN:E2 form, for the three month period between 1st January - 31st March 2007. Local research and development departments of each trust have also been contacted.

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff : Lead neonatologist for clinical governance in each maternity hospital in England.
* Babies born in England before 27 weeks gestation between January 2006 - 31st March 2007

Ages: 22 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Assess whether an innovative 'active' strategy for the dissemination of neonatal research findings, recs and national guidelines is more likely to lead to changes in policy and practice than the traditional,passive forms of dissemination in the UK. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Acolet, Principal Investigator — Confidential Enquiry into Maternal and Child Health